CLINICAL TRIAL: NCT03004560
Title: Psychology of Minimally Invasive Surgical Scars
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Duke University (Other)
Collaborators: Teleflex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00075024
Record Dates: First submitted 2016-12-20; First posted 2016-12-29 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Obesity
Keywords: Bariatric; standard laparoscopic surgery; minimally invasive; scars; psychology
MeSH Terms: conditions — Obesity; Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Laparoscopic Approach (Active Comparator): Minimally invasive laparoscopic procedure with 5-10 mm incisions.
  Interventions: Procedure: Standard Laparoscopic Approach
- Percutaneous Approach (Active Comparator): Minimally invasive laparoscopic procedure with 2-3 mm incisions.
  Interventions: Procedure: Percutaneous Approach

INTERVENTIONS:
Procedure: Standard Laparoscopic Approach — Minimally invasive laparoscopic surgery with 5-10 mm incisions.
  Arms: Standard Laparoscopic Approach
Procedure: Percutaneous Approach — Minimally invasive laparoscopic surgery with 2-3 mm incisions.
  Arms: Percutaneous Approach

SUMMARY:
The purpose of this study is to examine the psychological and psychosocial impact of surgical scars after minimally invasive surgery (MIS). 100 adult patients who are about to undergo bariatric procedures through the Duke Metabolic & Weight Loss Surgery program will be enrolled in this study. 50 patients will be randomly assigned to standard laparoscopic surgery and 50 will be assigned to the percutaneous group. All patients will complete pre-operative psychometric testing to establish a baseline body-image score as well as a patient's initial subjective perceptions around surgery and surgical scars. Follow-up visits will be done at standard of care timepoints - 3 weeks, 3 and 6 months, and 1 year after surgery. Subjects will complete the same psychometric measures to identify differences in psychological and psychosocial responses to standard laparoscopic and percutaneous scars. Patients will also complete a measure on scar satisfaction. The investigators hope to identify any differences between standard laparoscopic versus percutaneous approaches.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index 35 to 45
* Undergoing Bariatric Surgery

Exclusion Criteria:

* Body Mass Index <35 or >45
* Previous Bariatric Surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Scar satisfaction | Baseline, 3 weeks, 3 months, 6 months and 1 year post-op
  Patients will complete a scar assessment at post-op and routine follow up visits at 3 weeks, 3 months, 6 months, and 1 year.

SECONDARY OUTCOMES:
Change in the Abdominal pain scale | Baseline, 1 day post-op, 3 weeks, 3 months, 6 months and 1 year post-op
  Patients will complete an abdominal pain scale (0-10) at post-op and routine follow up visits at 3 weeks, 3 months, 6 months, and 1 year.

OTHER OUTCOMES:
Change in Psychometric testing questionnaire | Baseline, 3 weeks, 3 months, 6 months and 1 year post-op
  Psychometric testing will be performed to obtain a body image score and to see how/if that changes over time.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Portenier, MD, Principal Investigator — Duke University
Locations (1):
- Duke Center for Metabolic and Weight Loss Surgery, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No